CLINICAL TRIAL: NCT05104645
Title: Analysis of the Psychometric Properties of Kinematic Parameters of Locomotion Measured by Inertial Units. Validation in Healthy Volunteers and Stroke Patients
Acronym: KAPP-IMU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ORNETTI DIGITSOLE 2021
Record Dates: First submitted 2021-09-27; First posted 2021-11-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Vascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients after a Stroke (Experimental)
  Interventions: Other: Analysis of the walk
- Healthy Volunteering (Active Comparator)
  Interventions: Other: Analysis of the walk; Other: Analysis of the race; Other: Unipodal and bipodal jumps on flat ground

INTERVENTIONS:
Other: Analysis of the walk — Gait analysis in 3 dimensions and with inertial measurement units (IMUs) on flat ground and motorized treadmill Patients: S0, S1, S2, S4 and S6 Healthy volunteers: 2 times (between 3 and 20 days apart)
Other: Analysis of the race — Analysis of running in 3 dimensions and with inertial measurement units (IMUs) on flat ground and motorized treadmill Healthy volunteers: 2 times (between 3 and 20 days apart)
  Arms: Healthy Volunteering
Other: Unipodal and bipodal jumps on flat ground — Healthy volunteers: 2 times (between 3 and 20 days apart)
  Arms: Healthy Volunteering

SUMMARY:
Stroke is the leading cause of acquired disability in adults in France, and more than 500,000 French people are currently living with the after-effects. Hemiparesis, which is a partial deficit of motor or muscular control affecting the right or left half of the body, is the most frequent motor disorder after a stroke. Currently, the management and treatment of stroke patients consists of a combination of pharmacological treatments (drugs, botulinum toxin, etc.), the fitting of devices (orthoses, etc.) and rehabilitation (physical therapy, adapted physical activity, occupational therapy, etc.). According to the French National Authority for Health, motor rehabilitation after a stroke must meet 3 criteria: early, intensive and continuous. Functional evaluations (with validated measurement scales or analysis of locomotor activities) make it possible to monitor rehabilitation and to verify that the intensity is adapted to the patient's needs. To date, technological advances have yielded numerous gait analysis devices, ranging from motion capture platforms to inertial measurement units (IMU) and the use of motion platforms with integrated sensors. Different systems embedding an IMU on the foot, for example, answer these problems of analysis of walking in real situation. The IMUs record the movements and orientation of the foot in space; the data are then processed by algorithms to recognize the walking steps and calculate the spatiotemporal locomotion parameters. Additional IMUs positioned on the body can be added to this system in order to access a more precise analysis of locomotion, in particular by calculating the movements of the various joints of the lower limb. The validation of systems integrating IMUs must be done according to a precise method widely documented by the COSMIN recommendations (COnsensus-based Standards for the selection of health Measurement INstruments). This project will be carried out in two stages, the first of which will evaluate the safety and psychometric properties of the spatiotemporal parameters of the IMU devices in healthy subjects. If these properties (safety, reproducibility and validity) are considered to be in conformity, the second phase will be initiated. These same parameters will be evaluated during the rehabilitation of a cohort of patients who have suffered a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:
* Person who has given oral consent
* man or woman 18 years or older
* a person who is able to understand simple orders, instructions for locomotion
* person living within a maximum radius of 50 km from the investigation site

Patients (in addition to the above):

* persons who have had a stroke of any origin in the last 6 months
* person included in a rehabilitation protocol

Exclusion Criteria:

* persons who are not affiliated to national health insurance
* persons subject to a legal protection measure (guardianship)
* persons who are subject to a legal protection measure
* pregnant women
* adult unable to express consent
* subject with a disarticulated hip
* Subjects with diseases or disabilities that have an impact on walking other than those related to the stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Patients: Change from baseline at week 6
Walking speed | Healthy volunteers: Change from baseline at 20 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France